CLINICAL TRIAL: NCT03382262
Title: A Randomized, Open-label Study Comparing the Systemic Exposure to Triamcinolone Acetonide Following a Single Intra-articular Dose of Extended-release FX006 or Immediate-release TAcs (Triamcinolone Acetonide Suspension) in Patients With Osteoarthritis of the Shoulder (Glenohumeral Joint) or Hip
Brief Title: Study to Compare Exposure of TA Following Administration of FX006 or TAcs in Patients With OA of the Shoulder or Hip
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FX006-2017-013
Record Dates: First submitted 2017-12-06; First posted 2017-12-22 (Actual); Results first posted 2019-12-09 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Shoulder; Osteoarthritis of the Hip
Keywords: Osteoarthritis; Shoulder; Hip; Pain; Intra-articular; Injection; Corticosteroid
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis; Pain | interventions — FX006; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FX006 32 mg (Experimental): Single intra-articular (IA) injection of FX006 32 mg
  Interventions: Drug: FX006 32 mg
- TAcs 40 mg (Active Comparator): Single intra-articular (IA) injection of TAcs 40 mg
  Interventions: Drug: TAcs 40 mg

INTERVENTIONS:
Drug: FX006 32 mg — Extended-release 32 mg FX006 IA injection
  Other Names: Zilretta
  Arms: FX006 32 mg
Drug: TAcs 40 mg — Immediate-release 40mg TAcs IA injection
  Other Names: Kenalog®-40 Injection; Triamcinolone Acetonide Crystalline Suspension (TAcs); TCA-IR 40
  Arms: TAcs 40 mg

SUMMARY:
This is an open-label study to compare systemic exposure to triamcinolone acetonide following a dose of extended-release FX006 or immediate-release TAcs (triamcinolone acetonide suspension) in patients with osteoarthritis of the shoulder (glenohumeral joint) or hip

DETAILED DESCRIPTION:
This is a randomized, open-label, single dose study that will be conducted in male and female patients ≥40 years of age with OA of either the shoulder or the hip.

Approximately 24 patients with OA of the shoulder and approximately 24 patients with OA of the hip will be randomized to one of two treatment groups (1:1) and treated with a single IA injection of either:

* 32 mg FX006 (approximately 12 patients per joint) or
* 40 mg TAcs (approximately 12 patients per joint)

Each patient will be screened to confirm the diagnosis of OA of either the shoulder or hip and eligibility based on the other inclusion/exclusion requirements and will be randomized to treatment on Day 1. Each patient will be evaluated for a total of 12 weeks following the IA injection. Following screening, sampling for pharmacokinetics (PK) and safety will be completed at 10 out-patient visits scheduled on Study Days 1 [calendar day of injection], 2, 3, 5, 8, 15, 22, 29, 57, and 85.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Male or female greater than or equal to 40 years of age
* Body mass index (BMI) less than or equal to 40 kg/m2
* Ambulatory and in good general health
* Willing and able to comply with the study procedures and visit schedules and able to follow verbal and written instructions
* Willing to abstain from use of protocol-restricted treatments from Screening through End-of-Study visit
* Symptoms consistent with OA of the index joint for ≥ 6 months prior to Screening (patient reported is acceptable)
* Pain in the index joint for greater than15 days over the last month (as reported by the patient)
* For Shoulder OA patients: Radiologic findings of OA of the index shoulder meeting the Samilson-Prieto (S-P) Classification Grades 2 or 3
* For Hip OA patients: ACR Criteria (clinical and radiological) for OA of the index hip

Exclusion Criteria:

* Reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease
* History of infection in the index joint
* Clinical findings consistent with active infection or crystal disease in the index joint within 1 month of Screening
* History of fracture in the index limb within 12 months of Screening, or fracture with sequelae at any time
* Planned or anticipated surgery of the index joint during the study period
* Index joint instability or history of acute dislocation within 12 months of Screening
* If shoulder is the index joint, history of full or partial rotator cuff tear or significantly compromised rotator cuff function that, in the opinion for the Investigator, increases the difficulty or risk of IA injection
* Presence of surgical hardware or other foreign body in the index joint
* Surgery or arthroscopy of the index joint within 12 months of Screening
* IA treatment of any joint with any of the following agents within 6 months of Screening:
* Any corticosteroid preparation (investigational or marketed, including FX006), any biologic agent (e.g., platelet rich plasma (PRP) injection, stem cells, prolotherapy, amniotic fluid injection; investigational or marketed)
* IA treatment of the index joint with hyaluronic acid (investigational or marketed) within 6 months of Screening
* Parenteral or oral corticosteroids (investigational or marketed) within 3 months of Screening
* Inhaled, intranasal or topical corticosteroids (investigational or marketed) within 2 weeks of Screening
* Females who are pregnant or nursing or plan to become pregnant during the study; men who plan to conceive during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kelley, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (6):
- United States (6):
  - TriWest Research Associates, LLC, El Cajon, California
  - Biosolutions Clinical Research Center, La Mesa, California
  - Artemis Institute for Clinical Research, San Diego, California
  - LA Biomed at Harbor-UCLA Medical Center, Torrance, California
  - Rochester Clinical Research, Rochester, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

REFERENCES:
- [Derived] Kivitz A, Mehra P, Hanson P, Kwong L, Cinar A, Lufkin J, Kelley S. A Randomized, Open-Label, Single-Dose Study to Assess Safety and Systemic Exposure of Triamcinolone Acetonide Extended-Release in Patients With Hip Osteoarthritis. Rheumatol Ther. 2022 Apr;9(2):679-691. doi: 10.1007/s40744-022-00430-3. Epub 2022 Mar 8. PMID 35258839
- [Derived] Hanson P, Kivitz A, Mehra P, Kwong L, Cinar A, Lufkin J, Kelley SD. Safety and Systemic Exposure of Triamcinolone Acetonide Following Ultrasound-Guided Intra-Articular Injection of Triamcinolone Extended-Release or Standard Triamcinolone Acetonide in Patients with Shoulder Osteoarthritis: An Open-Label, Randomized Study. Drugs R D. 2021 Sep;21(3):285-293. doi: 10.1007/s40268-021-00348-1. Epub 2021 Aug 4. PMID 34350546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study was from December 2017 to July 2018. The patients were enrolled at medical clinics.
Groups:
- FX006 32 mg Shoulder: Single intra-articular (IA) injection of FX006 32 mg
  FX006 32 mg: Extended-release 32 mg FX006 IA injection in the Shoulder
- TAcs 40 mg Shoulder: Single intra-articular (IA) injection of TAcs 40 mg
  TAcs 40 mg: Immediate-release 40mg TAcs IA injection in the Shoulder
- FX006 32 mg Hip: Single intra-articular (IA) injection of FX006 32 mg
  FX006 32 mg: Extended-release 32 mg FX006 IA injection in the Hip
- TAcs 40 mg Hip: Single intra-articular (IA) injection of TAcs 40 mg
  TAcs 40 mg: Immediate-release 40mg TAcs IA injection in the Hip
Period: Overall Study
Arm/Group | FX006 32 mg Shoulder | TAcs 40 mg Shoulder | FX006 32 mg Hip | TAcs 40 mg Hip
Started | 12 | 13 | 15 | 15
Completed | 12 | 13 | 14 | 14
Not Completed | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FX006 32 mg Shoulder: Single intra-articular (IA) injection of FX006 32 mg in the Shoulder
  FX006 32 mg: Extended-release 32 mg FX006 IA injection
- TAcs 40 mg Shoulder: Single intra-articular (IA) injection of TAcs 40 mg in the Shoulder
  TAcs 40 mg: Immediate-release 40mg TAcs IA injection
- FX006 32 mg Hip: Single intra-articular (IA) injection of FX006 32 mg in the Hip
  FX006 32 mg: Extended-release 32 mg FX006 IA injection
- TAcs 40 mg Hip: Single intra-articular (IA) injection of TAcs 40 mg in the Hip
  TAcs 40 mg: Immediate-release 40mg TAcs IA injection
- Total: Total of all reporting groups
Arm/Group | FX006 32 mg Shoulder | TAcs 40 mg Shoulder | FX006 32 mg Hip | TAcs 40 mg Hip | Total
Number analyzed (Participants) | 12 | 13 | 15 | 15 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Consent
  years | 63.2 (11.39) | 61.9 (8.10) | 58.1 (7.60) | 60.1 (7.09) | 60.7 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 8 | 5 | 28
  Male | 3 | 7 | 7 | 10 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 1 | 1 | 5
  Not Hispanic or Latino | 9 | 13 | 14 | 14 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 2 | 5 | 5 | 13
  White | 10 | 11 | 8 | 9 | 38
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 15 | 15 | 55
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/mg^2] — Body Mass Index calculated at Baseline
  kg/mg^2 | 28.9 (5.98) | 30.7 (3.59) | 29.3 (3.49) | 31.0 (4.40) | 30.01 (4.367)

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Triamcinolone Acetonide (TA) in Blood Plasma
Description: Characterize the Pharmacokinetic Profile of FX006 and TCA IR [Time Frame: Day 1 (pre-treatment,1, 2, 3, 4, 5, 6, 8,10, and 12 hrs. post-dose) and Days 2, 3, 5, 8, 15, 22, 29, 57,and 85]
  For the PK analysis and individual concentration vs. time plots, a concentration that is BLOQ is assigned a value of zero if it occurs in a profile before the first measurable concentration. If a BLOQ value occurs after a measurable concentration in a profile and is followed by a value above the lower limit of quantification, then the BLOQ is treated as missing data. If a BLOQ value occurs at the end of the collection interval (after the last quantifiable concentration) it is set to zero. If two BLOQ values occur in succession after Cmax, the profile is deemed to have terminated at the first BLOQ value and any subsequent concentrations are set to zero for PK calculations
Time Frame: 12 Weeks
Population: All patients in the Safety population who received study drug, completed scheduled sampling and had sufficient plasma concentration data. 50 of 55 patients were included. Four unique patients for whom hip was the index joint were excluded due to IP administration deviations. One of the four was also found to be enrolled at 2 separate study centers.
Measure: Geometric Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | FX006 32 mg Shoulder | TAcs 40 mg Shoulder | FX006 32 mg Hip | TAcs 40 mg Hip
Number analyzed (Participants) | 12 | 13 | 11 | 14
pg/mL
  Day 1 - Hour 1 | 1061.8 [819.95 to 1375.09] | 1104.1 [578.17 to 2108.52] | 681.8 [334.47 to 1389.69] | 3862.3 [2024.11 to 7370.02]
  Day 1 - Hour 2 | 1117.6 [838.98 to 1488.62] | 1344.8 [682.40 to 2650.05] | 752.2 [364.55 to 1551.90] | 4052.4 [2134.61 to 7693.33]
  Day 1 - Hour 3 | 1140.0 [849.77 to 1529.44] | 1501.8 [774.05 to 2913.69] | 748.0 [349.37 to 1601.44] | 4519.3 [2286.88 to 8930.88]
  Day 1 - Hour 4 | 1142.4 [822.55 to 1586.49] | 1594.1 [856.43 to 2967.05] | 776.1 [352.73 to 1707.82] | 4557.8 [2362.49 to 8793.00]
  Day 1 - Hour 5 | 1093.8 [759.94 to 1574.40] | 1662.7 [861.73 to 3208.09] | 792.9 [360.39 to 1744.51] | 4672.6 [2429.24 to 8987.65]
  Day 1 - Hour 6 | 1052.8 [729.94 to 1518.37] | 1689.6 [893.53 to 3194.85] | 743.5 [331.07 to 1669.73] | 4469.8 [2393.87 to 8346.03]
  Day 1 - Hour 8 | 1016.2 [702.66 to 1469.64] | 1668.3 [887.88 to 3134.86] | 705.0 [307.07 to 1618.77] | 4102.3 [2232.93 to 7536.76]
  Day 1 - Hour 10 | 951.4 [670.78 to 1349.34] | 1506.3 [819.27 to 2769.61] | 698.2 [307.74 to 1583.97] | 3615.6 [2033.96 to 6427.30]
  Day 1 - Hour 12: number analyzed (Participants) | 10 | 13 | 11 | 14
  Day 1 - Hour 12 | 903.8 [637.58 to 1281.10] | 1531.3 [806.98 to 2905.65] | 675.1 [296.00 to 1539.62] | 3276.2 [1858.64 to 5775.00]
  Day 2 - Hour 24 | 943.4 [690.74 to 1288.35] | 1467.0 [884.10 to 2434.35] | 791.0 [340.46 to 1837.60] | 3218.8 [1965.24 to 5272.05]
  Day - 3 | 903.4 [639.75 to 1275.69] | 1413.1 [856.25 to 2332.05] | 682.1 [292.51 to 1590.60] | 1723.6 [1218.72 to 2437.70]
  Day - 5: number analyzed (Participants) | 11 | 13 | 11 | 14
  Day - 5 | 754.6 [536.22 to 1061.93] | 1038.2 [724.11 to 1488.44] | 562.4 [242.23 to 1305.93] | 897.3 [644.77 to 1248.66]
  Day - 8 | 678.1 [497.82 to 923.66] | 857.8 [596.48 to 1233.52] | 472.3 [202.04 to 1103.90] | 525.3 [296.03 to 932.01]
  Day - 15: number analyzed (Participants) | 12 | 12 | 10 | 14
  Day - 15 | 397.6 [287.43 to 549.88] | 722.7 [574.45 to 909.25] | 382.6 [270.89 to 540.52] | 444.7 [278.24 to 710.85]
  Day - 22 | 268.3 [186.53 to 385.82] | 476.7 [333.94 to 680.44] | 235.0 [170.80 to 323.29] | 331.6 [214.93 to 511.48]
  Day - 29 | 201.0 [134.57 to 300.21] | 418.7 [300.39 to 583.66] | 256.3 [173.31 to 379.15] | 281.8 [179.32 to 442.91]
  Day - 57: number analyzed (Participants) | 12 | 13 | 11 | 13
  Day - 57 | 151.8 [92.60 to 248.73] | 200 [140.83 to 284.08] | 225.1 [156.31 to 324.15] | 133.1 [74.28 to 238.50]
  Day - 85 | 100.1 [54.22 to 184.86] | 131.4 [64.14 to 269.25] | 112.0 [58.14 to 215.61] | 92.5 [51.16 to 167.11]

2. Primary Outcome: Total Number of Treatment Emergent Adverse Events
Description: Analyses of adverse events (AE) were performed for events considered treatment-emergent (TE). TE was defined as any AE with onset after administration of the 1st dose of study drug or any event present at baseline but worsened in intensity through the study. Severity was graded by the PI using the Common Terminology Criteria for AEs Version 4.0. Grading went from Grade 1 (Mild) to Grade 5 (Death Related to AE).
Time Frame: 12 Weeks
Population: All patients randomized to receive either FX006 or TAcs in the hip or shoulder.
Measure: Number; unit: Events
Arm/Group | FX006 32 mg Shoulder | TAcs 40 mg Shoulder | FX006 32 mg Hip | TAcs 40 mg Hip
Number analyzed (Participants) | 12 | 13 | 15 | 15
Events | 10 | 7 | 8 | 17

ADVERSE EVENTS:
Time Frame: Adverse events were collected following IA administration through the final study visit at 12 weeks.
Arm/Group | FX006 32 mg Shoulder | TAcs 40 mg Shoulder | FX006 32 mg Hip | TAcs 40 mg Hip
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 4/12 | 3/13 | 4/15 | 7/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32 mg Shoulder (N=12) | TAcs 40 mg Shoulder (N=13) | FX006 32 mg Hip (N=15) | TAcs 40 mg Hip (N=15)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Hypoaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — And Administrative Site Conditions
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular Pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic Hypoplasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
4 patients with hip as index joint, were excluded from the PK population. 3 patients had incomplete FX006 administration. 1 patient enrolled at 2 different study centers; receiving TAcs and FX006 5 days apart in the same hip with no TEAEs reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT03382262/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT03382262/SAP_001.pdf